CLINICAL TRIAL: NCT01437501
Title: Broccoli Sprout Intervention in Qidong, P.R. China
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Johns Hopkins University (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH); Qidong Liver Cancer Institute (Other); University of Pittsburgh (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00003494; 5P01ES006052 (NIH)
Record Dates: First submitted 2011-09-15; First posted 2011-09-21 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Environmental Carcinogenesis
Keywords: glucoraphanin; sulforaphane; pharmacokinetics; pharmacodynamics; broccoli sprout; carcinogens, environment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Broccoli Sprout Extract Beverage (Experimental)
  Interventions: Drug: Broccoli Sprout Extract Beverage
- Placebo beverage (Placebo Comparator)
  Interventions: Drug: placebo beverage

INTERVENTIONS:
Drug: Broccoli Sprout Extract Beverage — Broccoli Sprout Extract Beverage: 600 micromole glucoraphanin and 40 micromole sulforaphane dissolved in 100 mL dilute pineapple and lime juice daily for 84 days.
  Arms: Broccoli Sprout Extract Beverage
Drug: placebo beverage — 100 mL of dilute pineapple and lime juice daily for 84 days.
  Arms: Placebo beverage

SUMMARY:
This study is a 12 week placebo-controlled Phase II broccoli sprout intervention to be conducted in Qidong, P.R. China. One thousand two hundred people from the farming townships will be screened and three hundred eligible individuals will be enrolled in the study. Participants will be randomized into two treatment groups: one will receive a juice beverage containing glucoraphanin- and sulforaphane-rich broccoli sprout extract, pineapple juice, lime juice, and water and the other will receive a placebo beverage containing pineapple juice, lime juice and water. Participants will drink their assigned beverage every evening and provide biweekly urine samples and monthly blood samples. The principal endpoints of this study are pharmacokinetic evaluation of elimination of glucoraphanin/sulforaphane and their metabolites in urine and pharmacodynamic evaluation through measures of urinary levels of exposure biomarkers for dietary and air-borne toxins, which are known to be high in this population.

ELIGIBILITY:
Inclusion Criteria:

* age 21-65 years
* in good general health with no history of chronic illness
* normal liver function tests: alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin)
* normal renal function tests (creatinine, blood urea nitrogen, urinalysis)
* serum alpha-fetoprotein negative

Exclusion Criteria:

* personal history of cancer except for non-melanoma skin cancer
* use of prescribed medications
* hepatomegaly by clinical exam
* for women, a positive pregnancy test

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Kensler, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Qidong Liver Cancer Institute, Qidong, Jiangsu, China

REFERENCES:
- [Background] Kensler TW, Chen JG, Egner PA, Fahey JW, Jacobson LP, Stephenson KK, Ye L, Coady JL, Wang JB, Wu Y, Sun Y, Zhang QN, Zhang BC, Zhu YR, Qian GS, Carmella SG, Hecht SS, Benning L, Gange SJ, Groopman JD, Talalay P. Effects of glucosinolate-rich broccoli sprouts on urinary levels of aflatoxin-DNA adducts and phenanthrene tetraols in a randomized clinical trial in He Zuo township, Qidong, People's Republic of China. Cancer Epidemiol Biomarkers Prev. 2005 Nov;14(11 Pt 1):2605-13. doi: 10.1158/1055-9965.EPI-05-0368. PMID 16284385
- [Background] Egner PA, Chen JG, Wang JB, Wu Y, Sun Y, Lu JH, Zhu J, Zhang YH, Chen YS, Friesen MD, Jacobson LP, Munoz A, Ng D, Qian GS, Zhu YR, Chen TY, Botting NP, Zhang Q, Fahey JW, Talalay P, Groopman JD, Kensler TW. Bioavailability of Sulforaphane from two broccoli sprout beverages: results of a short-term, cross-over clinical trial in Qidong, China. Cancer Prev Res (Phila). 2011 Mar;4(3):384-95. doi: 10.1158/1940-6207.CAPR-10-0296. PMID 21372038

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1205 Individuals were recruited from HeHe Township in Qidong, PRC for eligibility screening at 3 medical clinics within the township in September 2011.
Groups:
- Broccoli Sprout Extract Beverage: Broccoli Sprout Extract Beverage : Broccoli Sprout Extract Beverage: 600 micromole glucoraphanin and 40 micromole sulforaphane dissolved in 100 mL dilute pineapple and lime juice daily for 84 days.
- Placebo Beverage: placebo beverage : 100 mL of dilute pineapple and lime juice daily for 84 days.
Period: Overall Study
Arm/Group | Broccoli Sprout Extract Beverage | Placebo Beverage
Started | 148 | 143
Completed | 135 | 132
Not Completed | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Broccoli Sprout Extract Beverage | Placebo Beverage | Total
Number analyzed (Participants) | 148 | 143 | 291
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 148 | 143 | 291
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (9.4) | 52.6 (7.7) | 51.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 111 | 229
  Male | 30 | 32 | 62
Region of Enrollment [Number; unit: participants]
  China | 148 | 143 | 291

OUTCOME MEASURES:

1. Primary Outcome: Effect of Treatment on Levels of Air Toxics Mercapturic Acids Over Intervention Period
Description: Urinary excretion of benzene mercapturic acid (S-PMA) in 12 hour overnight void at 12 weeks
Time Frame: Endpoints were assessed on urine samples collected at the end of the intervention on week 12.
Population: Analyses were conducted on all urine samples provided by study participants at week 12.
Measure: Median (Inter-Quartile Range); unit: pmol/mg creatinine
Arm/Group | Broccoli Sprout Extract Beverage | Placebo Beverage
Number analyzed (Participants) | 135 | 132
pmol/mg creatinine | 1.700 [1.235 to 2.386] | 1.065 [0.686 to 1.826]

2. Secondary Outcome: Levels of Sulforaphane and Its Metabolites at the End of Intervention Period (After 84 Daily Doses)
Description: Micromoles of urinary sulforaphane metabolites excreted over 24 hours after consuming the 84th dose.
Time Frame: Endpoints assessed on urine samples collected at the end of the intervention (day 84 [week 12])
Measure: Median (Inter-Quartile Range); unit: micromoles
Arm/Group | Placebo Beverage | Broccoli Sprout Extract Beverage
Number analyzed (Participants) | 132 | 135
micromoles | 1 [1 to 1] | 62 [44 to 91]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Broccoli Sprout Extract Beverage | Placebo Beverage
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/143
Other Adverse Events (participants affected / at risk) | 6/148 | 4/143
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Broccoli Sprout Extract Beverage (N=148) | Placebo Beverage (N=143)
light vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
indigestion (Gastrointestinal disorders) | 4 (4) | 2 (2)
taste (Gastrointestinal disorders) | 1 (1) | 2 (2) — participants disliked taste, worried about participation, withdrew from study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No